CLINICAL TRIAL: NCT06380387
Title: Whole Body Metabolism in Children Before and After Treatment of CNS Tumor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mette Cathrine Oerngreen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-21046543
Record Dates: First submitted 2024-02-21; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: CNS Tumor, Childhood
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meal intervention with stable isotopes (Experimental): A liquid mixed meal are gived adjusted by weight. The meal consists of: Intrinsically labelled D5-Phenylalanine and D3-Leucine labelled casein protein, 13C16palmitate, 13C6-Glucose in a mix of glucose, casein protein and rape seed oil dissolved in water in an energy density of 50% CHO, 35% fat and 15% protein. Blood samples are drawn frequently to measure fat, glucose and protein metabolism.
  Interventions: Dietary Supplement: Meal

INTERVENTIONS:
Dietary Supplement: Meal — Liquid meal

SUMMARY:
At the center of pediatric oncology in Copenhagen the investigators experience that the children with brain tumor, more or less have a healthy body with normal skeletal muscle mass and are physical active to the same level as their friends at the same age. The treatment period for brain tumor is approximately two years. After the treatment period, the children are more sedative with less interest in coming out doing physical activities and thus the investigators suspect that they have altered hormonal response, low skeletal muscle mass and perhaps are in risk of developing metabolic syndrome.

By comparing children with newly diagnosed CNS tumor with children finished treated for CNS tumor, we wish to describe the metabolic path during the approximately two years treatment period these children go through. These results will also be compared with results from healthy controls.

The investigators aim to include 10 children (aged 6-18 years) with newly diagnosed CNS tumor, 10 children (aged 6-18 years) finished treated for CNS tumor and 10 healthy controls (aged 6-18 years). By using stable isotope technique the investigators will investigate systemic fat, glucose and protein metabolism together with liver protein degradation and glucose production. Furthermore, by using DXA scan the investigators will describe the quality and distribution of skeletal muscle. Lastly, the investigators will determine the skeletal muscle signal pathway and metabolism in skeletal muscle via the Bergström biopsy technique in vastus lateralis.

DETAILED DESCRIPTION:
By comparing children with newly diagnosed CNS tumor with children finished treated for CNS tumor, the investigators wish to describe the metabolic path during the approximately two years treatment period these children go through. These results will also be compared with results from healthy controls.

Trial design and time frame:

A prospective, non-randomized, cross-sectional study.

There will be three different patient groups included:

* Patient group A: Children with newly diagnosed CNS tumor
* Patient group B: Children finished treated for CNS tumor
* Healthy controls: Children admitted to the hospital at the Epilepsy monitor unit (EMU)

The trial will be conducted over a total of two days and takes place at the Department of Pediatrics and Adolescent Medicine, Rigshospitalet and the Copenhagen Neuromuscular Center, Department of Neurology, Rigshospitalet.

* Study day 1: Is estimated to last approximately 2 hours.
* Study day 2: Is estimated to last approximately 8 hours.

Study Day 1: The children will be DXA-scanned and complete life quality questionnaires and pain scores. In some cases, study day 1 will be done after study day 2, depending on the cancer treatment plan for each patient.

Study Day 2: For the patients newly diagnosed with CNS tumor: The investigators strive to conduct study day 2 within the first week of hospital admission due to newly diagnosed CNS tumor. However, the investigators do accept study day 2 being conducted within the first month after time of diagnose.The subjects will arrive around 08.00, at Copenhagen Neuromuscular Centre (CNMC), Rigshospitalet.

On arrival, EMLA (local anesthetics cream) will be applied on the skin of the children in order to minimize any discomfort that may occur during iv-insertion. Two peripheral venous catheters are inserted, one in the medial cubital vein for infusion of stable isotopes, and one in a dorsal vein of the hand for blood sampling. If the child has a central venous catheter (CVK), we will only insert one peripheral venous catheter, in the medial cubital vein for infusion of the stable isotopes.

After 1 hour and 45 minutes of basal tracer infusion, basal blood samples are drawn (time -15 and 0) for the determination of basal steady state tracer enrichments and hormone concentrations. At time= 0, a liquid mixed meal is provided. Blood samples are drawn frequently for 6 hours relative to start of the test meal (at 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240, 300 and 360 minutes)[24], [25]. If the child becomes upset or we for other reasons want to stop earlier than 6 hours, we will use the already obtained results.

The tracers: In this study, the investigators will intravenously infuse small amounts of metabolites labelled with stable isotopes in primed continuous intravenous infusions of: D8-Phenylalanine, D2-Tyrosine, 13C18-Oleate acid, D2-Glucose, D5-Glycerol. This method is well-established at both CIMT and CNMC and has been used investigating several of patients categories before: Neonates (ongoing study), gastric sleeve, elderly and neuromuscular patients.

The tracers are prepared from the hospital pharmacy. All tracers are purchased from Cambridge Isotope Laboratories, Andover, MA, USA suitable for human use. Stable isotopes are non-radioactive and naturally occurring in food (e.g. in corn).

Food intervention: At time= 0 (120 minutes after infusion), a liquid mixed meal adjusted by weight is given. The meal consists of: Intrinsically labelled D5-Phenylalanine and D3-Leucine labelled casein protein, 13C16palmitate, 13C6-Glucose in a mix of glucose, casein protein and rape seed oil dissolved in water in an energy density of 50% CHO, 35% fat and 15% protein. Intrinsically labeled caseinate was produced via an infusion of [D5]-phenylalanine and [D3]leucine into a lactating cow to obtain enriched milk Foulumn, Arhus University, from which the caseinate fraction was isolated at Arla Foods according to Good Manufacturing Practice (GMP) and safety checked an store under appropriate regulatory conditions until use (Nørre Vium, Denmark) following a previously described procedure.

Analyses of blood samples:The samples will be collected in syringes containing 10μL EDTA/mL to prevent coagulation. The blood is immediately centrifuged at 4oC to separate plasma from red blood cells. The samples will be frozen in coded tubes and stored at -80C until analysis.

Routine blood samples: Will be analysed immediately at the Department of Clinical Biochemistry, Rigshospitalet:

- Blood samples include: Insulin, HbA1C, Cholesterol, HDL, LDL, triglycerides

Glucose and lactate: will be analyzed (ABL 700) immediately as the blood is drawn.

Specific blood samples:

* Free fatty acids: will be analyzed using fluorometry.
* Hormones (catecholamines, insulin, incretins and glucagon): will be analyzed using RIA and Elisa Methods respectively.
* Stable isotope enrichments in blood: will be analyzed using Liquid chromatography-tandem mass-spectrometry (LC-MS/MS) and gas chromatography combustion isotope ratio mass spectrometry (GC-C-IRMS) (Thermo Scientific, Palo Alto, CA, USA and Bremen, Germany).

Calculations: Whole body metabolite quantitative kinetics will be calculated using Steele's equation for non-steady state adapted for analysis of stable isotopes under the post-absorptive conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient group A: Children with newly diagnosed CNS tumor, included just before the start of treatment or right after possible surgery.
* Patient group B: Children who have completed treatment for a CNS tumor within the last month.
* Healthy controls: Children admitted to the EMU because of either

  * Suspected convulsions
  * Nocturnal EEG changes
* 6-18 years
* Signed informed consent to participation in the trial.

Exclusion Criteria:

* Inability to understand the purpose of the trial or cooperate in the conduction of the experiments. For the children this will concern of course the parents or the guardians of the child.
* Competing conditions at risk of compromising the results of the study.
* Participation in other trials that may interfere with the results.
* Intake of medications that may interfere with the results, evaluated by investigator.
* Pregnancy or breastfeeding.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Protein breakdown | 10 hours
  Phenylalanine Rate of appearance micro mol/kgFFM/min
Protein synthesis | 10 hours
  Phenylalanine Rate of disappearance micro mol/kgFFM/min
Phenylalanine concentration | 10 hours
  micromol/l
Phe oxidation to TYR | 10 hours
  micromol/kg FFM/min
Whole-body protein synthesis | 10 hours
  micromol Phe/kg FFM/min
Whole-body protein degradation | 10 hours
  micromol Phe /kg FFM/min
Netto protein balance | 10 hours
  micromol Phe /kg FFM/min
Glucose Rate of appearance | 10 hours
  micromol/kg FFM/min
Total glucose Rate of appearance | 10 hours
  micromol/kg FFM/min
Total glucose Rate of disappearance | 10 hours
  micromol/kg FFM/min
Endogenous glucose | 10 hours
  micromol/kg FFM/min
Oral phenylalanine Rate of appearance | 10 hours
  micromol/kg FFM/min
Phenylalanine oxidation | 10 hours
  % of phenylalanine Rate of appearance
Rate of Appearance of Palmitate in Plasma | 10 hours
  µmol/kg/min
Rate of Disappearance of Palmitate | 10 hours
  µmol/kg/min
Concentration of ketones | 10 hours
  mmol/L

SECONDARY OUTCOMES:
Glucose | 10 hours
  Nutritional, meal, absorption kinetics of proteins, carbohydrates and fat including first bypass losses (interstitial and liver). In case of fat that included synthesis rates of chylomicrons and their breakdown rate by determining the overflow of the nutritional fatty acids into the main circulation.
Quality of Skeletal Muscle | 10 hours
  Dual-energy X-ray absorptiometry (DEXA) scan
Protein synthesis rate | 10 hours
  Blood, mainly liver, proteins synthesis rate and liver function parameter from, A. liver glucose; B. VLDL-TAG production rate; C. phenylalanine hydroxylation rates
Pain score | 10 hours
  Pain score assessment (1-10)
Life quality score | 10 hours
  Life quality score by using PedsQL (0-100)
Muscle biopsy | 10 hours
  Muscle morphology, muscle fiber type and size, atrophy protein markers (MuRF1, MAFbx, FoxO) muscle generating markers (Myo D, Myogenin, IGF1), muscle growth regulating protein (myostatin).
Incretins | 10 hours
  GLP-1 (pmol/L) and GIP, (pmol/L)
Glucagon | 10 hours
  pmol/L
Liver parameters ALT, AST, GGT | 10 hours
  ALT, AST, GGT (U/L)
Bilirubin | 10 hours
  mikromol/L
International normalized ratio (INR) | 10 hours
  Blood sample
LDH | 10 hours
  U/L
Insulin | 10 hours
  pmol/L
catecholamines | 10 hours
  nmol/l nmol/l
Blood pressure | 10 hours
  mmHG
Waist- and hip circumference | 10 hours
  centimeter
Lipids | 10 hours
  HDL , LDL, total cholesterol, TAG (mmol/L)
Concentration of Plasma Amino Acids | 10 hours
  mmol/L
Concentration of Plasma Glucose | 10 hours
  mmol/L
Concentration of Plasma Palmitate | 10 hours
  micromol/L
Concentration of Plasma Free Fatty Acids | 10 hours
  mmol/L
Level of HbA1c | 10 hours
  mmol/mol

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics and Adolescent Medicine and Copenhagen Neuromuscular Center, Rigshospitalet, Copenhagen, Copenhagen Ø, Denmark

IPD SHARING:
Plan to Share IPD: No